CLINICAL TRIAL: NCT07360561
Title: Effect of Mobile Health-Based Gamified Long-Term Interventions to Increase Physical Activity on Cardiovascular Risk Factors
Brief Title: Effect of Mobile Health-Based Gamified Long-Term Interventions to Increase Physical Activity on Cardiovascular Risk Factors: Randomized Controlled Study on University Students and Employees
Acronym: mHealth Exerc
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ramiz ARABACI, Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-20/1; 324K201 (Other: TUBITAK 1002-A)
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Exercise; Physical Activity; Gamification; University Student; College Student
Keywords: exercise; physical activity; gamification; university student; college student
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of five parallel groups: walking intervention, gamified walking intervention, walking and exercise intervention, gamified walking and exercise intervention, or a no-intervention control group. All intervention groups will be followed concurrently for 12 weeks.
Who Masked: Participant
Masking Description: This study used single masking. Participants are blinded to the gamification component of the intervention and are not informed whether the walking and exercise program includes gamified elements. Due to the nature of the intervention, the researchers delivering it are aware of the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Walking intervention (WG) (Experimental): Participants will walk daily for 12 weeks to achieve a predetermined step goal.
  Interventions: Behavioral: Walking program
- Gamified walking intervention (GWG) (Experimental): Participants will walk daily for 12 weeks to achieve a predetermined step goal and will use a gamified application to support their walking.
  Interventions: Behavioral: Walking program; Behavioral: Gamified Mobile Application
- Walking and exercise intervention (WEG) (Experimental): Participants will walk daily for 12 weeks to achieve a predetermined step goal, perform high-intensity circuit training (HICT) for at least 15 minutes on three designated days per week.
  Interventions: Behavioral: Walking program; Behavioral: High-intensity circuit training (HICT)
- Gamified walking and exercise intervention (GWEG) (Experimental): Participants will walk daily for 12 weeks to achieve a predetermined step goal, perform high-intensity circuit training (HICT) for at least 15 minutes on three designated days per week, and use a gamified application to support walking and exercise activities.
  Interventions: Behavioral: Walking program; Behavioral: High-intensity circuit training (HICT); Behavioral: Gamified Mobile Application
- Control group (CG) (No Intervention): Participants will not receive any structured physical activity intervention and will continue their usual daily lifestyle throughout the study period.

INTERVENTIONS:
Behavioral: Walking program — Walk daily for 12 weeks to achieve a predetermined step goal.
  Arms: Gamified walking and exercise intervention (GWEG); Gamified walking intervention (GWG); Walking and exercise intervention (WEG); Walking intervention (WG)
Behavioral: High-intensity circuit training (HICT) — High-intensity circuit training performed for at least 15 minutes on three designated days per week for 12 weeks, in addition to daily walking.
  Arms: Gamified walking and exercise intervention (GWEG); Walking and exercise intervention (WEG)
Behavioral: Gamified Mobile Application — Use of a gamified application designed to promote motivation, adherence, and engagement in walking and exercise activities during the 12-week intervention period.
  Arms: Gamified walking and exercise intervention (GWEG); Gamified walking intervention (GWG)

SUMMARY:
The increasing incidence of cardiovascular disease (CVD) and related mortality is now recognized as a global emergency. CVD risk factors include unhealthy diet, inactivity, dyslipidemia, diabetes, high blood pressure, obesity, smoking, and family history/genetics. Increasing physical activity (PA) is recognized as an essential factor in reducing the risk of CVD. Many studies have emphasized that regular and adequate physical activity significantly reduces the risk of CVD through effects such as lowering blood pressure and cholesterol levels, supporting weight control, and improving diabetes management. Measuring steps/day is used to determine PA, and as technologies have developed, smartphones have become widely used tools. Inactivity and time constraints of modern life make it difficult for people to increase PA levels. Therefore, innovative intervention methods based on mobile health and gamification should be used to improve individuals' physical activity. Gamification is the application of game design elements such as points, badges, leaderboards, and levels in non-game environments. Gamification is increasingly being used to create change, particularly in physical activity and health behaviors. It is recommended to include resistance exercises at least 2 days a week in addition to aerobic activity to maximize health benefits. Recently, the high-intensity circuit training (HICT) program, which combines high-intensity interval training (HIIT) and circuit training (CT), requires less time, combines aerobic and resistance exercises, and uses body weight, has been developed and is used in sports. The main aim of the present study is to examine the effects of 12-week Mobile Health-Based Gamified applications on cardiovascular risk factors among university students and employees. In this direction, it is aimed to increase participants' daily steps and improve their physical activity habits. A total of 105 volunteers aged 18 to 64, including students and employees of Bursa Uludag University, will participate in the study. PACER pedometer and 7 Minute Workout HICT exercise mobile health applications will be used in the study.

Subjects will be divided into five equal groups of 21 people each using the closed opaque envelope randomization method. Walking intervention (WG), gamified walking intervention (GWG), walking and exercise intervention (WEG), gamified walking and exercise intervention (GWEG), and control (CG) groups will be formed. The first four groups (WG, GWG, WEG, and GWEG) will walk every day for 12 weeks to reach the set target number of steps. In addition, volunteers in the GWEG and WEG group will exercise (HICT) for at least 15 minutes on 3 designated days per week in addition to walking. In addition, volunteers in the GWG and GWEG groups will use a gamified application. In CG, there will be no regular physical activity, and they will continue their daily lifestyle. In our study, unlike those conducted to date, the application of HICT with gradually increasing physical activity for 12 weeks to reduce CVD risk factors, and the use of gamified methods to stay in the program and ensure sustainability, emphasize its unique value. The gamified exercise program applied in this study is expected to provide an additional benefit for CVD risk factors compared with the protocols used to date.

ELIGIBILITY:
Inclusion Criteria:

* Being among 18 or 65
* To give verbal and written consent to participate in the study voluntarily

Exclusion Criteria:

* If there are any health issues
* IPAQ>= 3000 MET / day (IPAQ: International Physical Activity Questionnaire - Short Form)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Body Composition and Anthropometric Measurements | From enrollment to the end of treatment at 12 weeks
  Body composition parameters will be assessed in study participants. Body weight (kg) and body fat percentage will be measured using the TANITA BC 418 MA device via bioelectrical impedance analysis. Waist and hip circumference measurements will be obtained using a measuring tape with 1 mm precision while participants are standing upright on a flat surface. Waist circumference will be measured at the level of the umbilicus, and hip circumference will be measured at the widest part of the hips by wrapping the measuring tape completely around the body. Body mass index (BMI) will be calculated by dividing body weight (kg) by the square of height (m²).
Cardiovascular Disease Risk Factors | From enrollment to the end of treatment at 12 weeks
  Cardiovascular disease (CVD) risk factors will be assessed according to the criteria defined by the American College of Sports Medicine (ACSM). Blood biochemical parameters, including total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, triglycerides, and fasting blood glucose, will be analyzed at the university hospital laboratory where the study is conducted. Systolic and diastolic blood pressure will be measured using an automated blood pressure monitor (Omron M2 Intellisense). Blood pressure will be measured in the right arm and repeated 3 times, with the mean used for analysis.
Physical Activity Level Assessed by the International Physical Activity Questionnaire-Short Form (IPAQ-SF) | From enrollment to the end of treatment at 12 weeks
  Participants' physical activity levels will be assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF), which is designed for individuals aged 15 to 65 years. The IPAQ-SF consists of seven items that assess the frequency and duration of walking, moderate-intensity physical activity, and vigorous-intensity physical activity over the previous 7 days.

SECONDARY OUTCOMES:
Daily Step Count Monitored via Google Fit | From enrollment to the end of treatment at 12 weeks
  Participants' daily step counts will be monitored using the Google Fit mobile application over 3 months. The intervention aims to increase the average daily step count during the monitoring period. Step count data recorded by Google Fit will be used for analysis.
Exercise Adherence to High-Intensity Circuit Training (HICT) via the "7 Minute Workout" Mobile Application | From enrollment to the end of treatment at 12 weeks
  Exercise participation will be monitored using the "7 Minute Workout" mobile application. Participants will be instructed to perform high-intensity circuit training (HICT) exercises at least three days per week. The HICT protocol consists of 12 high-intensity, bodyweight-based exercises and is evidence-based and supported by the American College of Sports Medicine (ACSM). Exercise adherence will be evaluated based on application-recorded activity data.

CONTACTS AND LOCATIONS:
Locations (1):
- Uludağ University, Faculty of Spor Science Lab, Bursa, NİLÜFER, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethical issues